CLINICAL TRIAL: NCT02282670
Title: A Phase III Clinical Trial to Evaluate the Efficacy and Safety of DA-5204 and to Demonstrate the Non-inferiority of DA-5204 Compared With Stillen Tab. in Patients With Acute or Chronic Gastritis
Brief Title: A Study to Evaluate the Efficacy and Safety of DA-5204
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA5204_GR_III
Record Dates: First submitted 2014-10-28; First posted 2014-11-04 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Acute Gastritis; Chronic Gastritis
MeSH Terms: interventions — DA-5204; DA 9601

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DA-5204 (Experimental): DA-5204 administered two times daily for two weeks
  Interventions: Drug: DA-5204
- Stillen tab. (Active Comparator): Stillen tab. administered three times daily for two weeks
  Interventions: Drug: Stillen tab.

INTERVENTIONS:
Drug: DA-5204
  Arms: DA-5204
Drug: Stillen tab.
  Arms: Stillen tab.

SUMMARY:
This is a multicenter, active-controlled, randomized, double-blinded, paralleled group clinical study to evaluate the efficacy and safety of DA-5204 and to demonstrate the non-inferiority of DA-5204 compared with Stillen® tab. in patients with acute or chronic gastritis.

ELIGIBILITY:
Inclusion Criteria:

* Age is over 20 years old, under 75 years old, men or women
* Patients diagnosed with acute or chronic gastritis by gastroscopy
* Patients with one or more erosions found by gastroscopy
* Signed the informed consent forms

Exclusion Criteria:

* Patients who is impossible to receive gastroscopy
* Patients with peptic ulcer and gastroesophageal reflux disease
* Patients administered with prokinetics, H2 receptor antagonists, proton pump inhibitors, anticholinergic drugs or non-steroid anti-inflammatory drugs prior to study in 2 weeks
* Patients with surgery related to gastroesophageal
* Patients with Zollinger-Ellison syndrome
* Patients with any kind of malignant tumor
* Patients administered with anti-thrombotic drugs
* Patients with significant cardiovascular, pulmonary, heptic, renal, hemopoietic or endocrine system primary disease
* Patients with neuropsychiatric disorder, alcoholism, or drug abuse
* Patients taking other investigational drugs or participating in other clinical studies in 4 weeks.
* Women either pregnant or breast feeding

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
A percentage of subjects showed moderate or significant improvement of stomach erosions by the endoscopy. | 2 weeks
  The definition of "moderate improvement" is the subjects showed score changed from 4 to 1 or from 2 to 1. And, "significant improvement" means the subject showed score changed from 4 to 1 or from 3 to 1.
  [score 1(normal) : no erosion, score 2(mild) : 1-2 erosions, score 3(moderate) : 3-5 erosions, score 4(severe) : 6 or more erosions]

SECONDARY OUTCOMES:
A percentage of completely cured subject after a treatment | 2 weeks
  The definition of "completely cured" is the subjects with no erosions, in other words, 0 erosion found at stomach by the endoscopy.
A percentage of subjects showed morderate or significant improvement of gastric symptom rating scale. | 2 weeks
  The definition of "moderate improvement" is the subjects showed reduction ratio of score changed from 50% to 75%. And, "singnificant improvement" means the subjects showed reduction ratio of score changed 75% or more. Reduction ratio of score is calculated as [1-(total score of 7 days before termination of treatment)/(total score of 7 days before treatment)].

CONTACTS AND LOCATIONS:
Overall Officials: Dong Ho Lee, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital of Korea; Myung Gyu Choi, M.D., Ph.D., Principal Investigator — The Catholic University, Seoul St. Mary's Hospital of Korea; Sung Joon Lee, M.D., Ph.D., Principal Investigator — Kangwon National University Hospital of Korea; Sung Kuk Kim, M.D., Ph.D., Principal Investigator — Kyungbuk National University Hospital of Korea; Geun Am Song, M.D., Ph.D., Principal Investigator — Pusan National Universtiy Hospital of Korea; Poong Lyeol Lee, M.D., Ph.D., Principal Investigator — Samsung Medical Center of Korea; Hwoon Yong Jung, M.D., Ph.D., Principal Investigator — Asan Medical Center of Korea; Dae Hwan Kang, M.D., Ph.D., Principal Investigator — Pusan National University Yangsan Hospital of Korea; Yong Chan Lee, M.D., Ph.D., Principal Investigator — Yonsei University, Severance Hospital of Korea; Si Hyung Lee, M.D., Ph.D., Principal Investigator — Yeungnam University Hospital of Korea; Suck Chei Choi, M.D., Ph.D., Principal Investigator — Wonkwang University Hospital of Korea; Gi Nam Sim, M.D., Ph.D., Principal Investigator — Ewha Womans University Medical Center of Korea; Sang Young Seoul, M.D., Ph.D., Principal Investigator — Inje University Busan Paik Hospital of Korea; Jeong Seop Moon, M.D., Ph.D., Principal Investigator — Inje University Seoul Paik Hospital of Korea; Yong Woon Shin, M.D., Ph.D., Principal Investigator — Inha University Hospital of Korea; Hyen Soo Kim, M.D., Ph.D., Principal Investigator — Chonnam National Universtiy Hospital of Korea; Soo Teik Lee, M.D., Ph.D., Principal Investigator — Chonbuk National Universtiy Hospital of Korea; Jin Woong Cho, M.D., Ph.D., Principal Investigator — The Presbyterian medical center in Jeonju of Korea; Eun Kwang Choi, M.D., Ph.D., Principal Investigator — Jeju National Universtiy Hospital of Korea; Soon Man Yoon, M.D., Ph.D., Principal Investigator — Chungbuk National University Hospital of Korea; Oh Young Lee, M.D., Ph.D., Principal Investigator — Hanyang Universtiy Hospital of Korea; Jin Seok Jang, M.D., Ph.D., Principal Investigator — Dong-A University Hospital of Korea
Locations (1):
- Seoul National Universtiy, Bundang Hospital, IRB, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Choi YJ, Lee DH, Choi MG, Lee SJ, Kim SK, Song GA, Rhee PL, Jung HY, Kang DH, Lee YC, Lee SH, Choi SC, Shim KN, Seol SY, Moon JS, Shin YW, Kim HS, Lee ST, Cho JW, Choi EK, Lee OY, Jang JS. Evaluation of the Efficacy and Safety of DA-9601 versus Its New Formulation, DA-5204, in Patients with Gastritis: Phase III, Randomized, Double-Blind, Non-Inferiority Study. J Korean Med Sci. 2017 Nov;32(11):1807-1813. doi: 10.3346/jkms.2017.32.11.1807. PMID 28960033